CLINICAL TRIAL: NCT01463813
Title: Finnish Vitamin D Trial (FIND)
Acronym: FIND
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Eastern Finland (Other)
Collaborators: Academy of Finland (Other); Juho Vainio Foundation (Other); Finnish Foundation for Cardiovascular Research (Other); Finnish Cultural Foundation (Other)
Responsible Party: Principal Investigator, Tomi-Pekka Tuomainen, Professor, University of Eastern Finland
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: FIND
Record Dates: First submitted 2011-10-13; First posted 2011-11-02 (Estimated); Last update posted 2018-10-23 (Actual); Status verified 2018-10

CONDITIONS: Cardiovascular Diseases; Cancer
Keywords: bone density conservation agents; cancer; cardiovascular disease; cholecalciferol; diabetes mellitus, type 2; dietary supplements; primary prevention; vitamin D
MeSH Terms: conditions — Cardiovascular Diseases; Neoplasms; Diabetes Mellitus, Type 2 | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Placebo Comparator): Placebo, no Vitamin D3
  Interventions: Dietary Supplement: Placebo
- Vitamin D3 80 (Experimental): Vitamin D3 80 micrograms (3200 IU) per day
  Interventions: Dietary Supplement: Vitamin D3
- Vitamin D3 40 (Experimental): Vitamin D3 40 micrograms (1600 IU) per day
  Interventions: Dietary Supplement: Vitamin D3

INTERVENTIONS:
Dietary Supplement: Vitamin D3 — Vitamin D3 40 micrograms (1600 IU) per day
  Other Names: Cholecalciferol
  Arms: Vitamin D3 40
Dietary Supplement: Vitamin D3 — Vitamin D3 80 micrograms (3200 IU) per day
  Other Names: Cholecalciferol
  Arms: Vitamin D3 80
Dietary Supplement: Placebo — Inactive placebo
  Arms: Placebo

SUMMARY:
The Finnish Vitamin D Trial (FIND) is a randomized, double-blind, placebo-controlled, 5-year supplementation study of the benefits and risks of vitamin D in the primary prevention of cardiovascular (CVD) and cancer among 18000 men 60 years or older and women 65 years or older.

[Edit 25.3.2015: Due to difficulties in recruitment and funding, the study size is approximately 2500 subjects, with a 550 subject subgroup with more detailed examinations]

The participants will be randomized to 3 groups with 6000 in each, with daily supplementation of either: 1) 40 µg/day (1600 IU) of vitamin D3, 2) 80 µg/day (3200 IU) of vitamin D3, or 3) placebo.

[Edit 15.3.2015: The 2500 subjects are randomized in 3 groups, approximately 830 subjects per group.]

Compliance, use of non-study drugs or supplements, diet, development of endpoints, and CVD and cancer risk factors will be assessed by questionnaires. Blood samples will be collected for assessment of effect modification by baseline 25-hydroxyvitamin D, as well as for future ancillary studies of genetic/biochemical hypotheses. Event data will be obtained by record linkage from the national computerized hospitalization registry.

DETAILED DESCRIPTION:
More detailed description available upon request.

ELIGIBILITY:
Inclusion Criteria:

* Men 60 years or older
* Women 65 years or older

Exclusion Criteria:

* Cardiovascular disease (including myocardial infarction, stroke, transient ischemic attack, angina pectoris, coronary artery bypass grafting, or percutaneous coronary intervention).
* Cancer (except non-melanoma skin cancer).
* Any disease or state that raises a vitamin D related safety concern (such as chronic liver, thyroid or kidney disease, hypercalcemia, sarcoidosis or other granulomatous diseases such as active chronic tuberculosis or Wegener's granulomatosis).
* Use of supplements yielding vitamin D over 20 µg/day or calcium over 1200 mg/day and unwillingness to discontinue the use.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2495 (Actual)
Dates: Start 2012-09 (Actual); Primary Completion 2018-10 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Cardiovascular disease | 5 years
  CVD incidence in VitD arms vs. placebo arm.
Cancer | 5 years
  Cancer incidence in VitD arms vs.placebo arm

CONTACTS AND LOCATIONS:
Overall Officials: Tomi-Pekka Tuomainen, MD, PhD, Principal Investigator — University of Eastern Finland; Jyrki K Virtanen, PhD, Principal Investigator — University of Eastern Finland; Sari Voutilainen, PhD, Principal Investigator — University of Eastern Finland
Locations (1):
- University of Eastern Finland, Kuopio Campus, Kuopio, Northern Savonia, Finland

REFERENCES:
- [Derived] Rikkonen T, Hantunen S, Kroger H, Lamberg-Allardt C, Manson JE, Nurmi T, Tuppurainen M, Voutilainen A, Tuomainen TP, Virtanen JK. The Effect of Vitamin D3 Supplementation on the Risk of Falls in a General Population-The Finnish Vitamin D Trial. J Am Geriatr Soc. 2026 Jan 13. doi: 10.1111/jgs.70295. Online ahead of print. PMID 41531181
- [Derived] Ahl NM, Hantunen S, Tuomainen TP, Lamberg-Allardt C, Manson JE, Nurmi T, Uusitupa M, Voutilainen A, Tolmunen T, Virtanen JK. Vitamin D supplementation and incidence of major depressive disorder - A randomized clinical trial. Clin Nutr. 2026 Feb;57:106570. doi: 10.1016/j.clnu.2025.106570. Epub 2025 Dec 30. PMID 41506003
- [Derived] Lonnroos E, Ylilauri M, Lamberg-Allardt C, Manson JE, Nurmi T, Uusitupa M, Voutilainen A, Hantunen S, Tuomainen TP, Virtanen JK. The Effect of Vitamin D3 Supplementation on the Incidence of Diagnosed Dementia Among Healthy Older Adults-The Finnish Vitamin D Trial. J Gerontol A Biol Sci Med Sci. 2025 Jun 10;80(7):glaf077. doi: 10.1093/gerona/glaf077. PMID 40243375
- [Derived] Virtanen JK, Hantunen S, Kallio N, Lamberg-Allardt C, Manson JE, Nurmi T, Pihlajamaki J, Uusitupa M, Voutilainen A, Tuomainen TP. The effect of vitamin D3 supplementation on the incidence of type 2 diabetes in healthy older adults not at high risk for diabetes (FIND): a randomised controlled trial. Diabetologia. 2025 Apr;68(4):715-726. doi: 10.1007/s00125-024-06336-9. Epub 2024 Dec 2. PMID 39621103
- [Derived] Virtanen JK, Hantunen S, Lamberg-Allardt C, Manson JE, Nurmi T, Uusitupa M, Voutilainen A, Tuomainen TP. The effect of vitamin D3 supplementation on atrial fibrillation in generally healthy men and women: The Finnish Vitamin D Trial. Am Heart J. 2023 Oct;264:177-182. doi: 10.1016/j.ahj.2023.05.024. Epub 2023 Jun 10. PMID 37302737